CLINICAL TRIAL: NCT02718417
Title: A RANDOMIZED, OPEN-LABEL, MULTICENTER, PHASE 3 STUDY TO EVALUATE THE EFFICACY AND SAFETY OF AVELUMAB (MSB0010718C) IN COMBINATION WITH AND/OR FOLLOWING CHEMOTHERAPY IN PATIENTS WITH PREVIOUSLY UNTREATED EPITHELIAL OVARIAN CANCER JAVELIN OVARIAN 100
Brief Title: Avelumab in Previously Untreated Patients With Epithelial Ovarian Cancer (JAVELIN OVARIAN 100)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated based on the results of a planned interim analysis that showed futility of efficacy.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B9991010; 2015-003239-36 (EudraCT Number); JAVELIN OVARIAN 100 (Other: Alias Study Number)
Record Dates: First submitted 2016-03-15; First posted 2016-03-24 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Ovarian Cancer
Keywords: untreated epithelial ovarian; fallopian tube; primary peritoneal cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; Paclitaxel; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Active Comparator): Chemotherapy followed by observation
  Interventions: Drug: carboplatin; Drug: paclitaxel
- Arm B (Experimental): Chemotherapy followed by avelumab in maintenance
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: Avelumab
- Arm C (Experimental): Chemotherapy in combination with avelumab followed by avelumab in maintenance
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: Avelumab

INTERVENTIONS:
Drug: carboplatin — Given Q3W during chemotherapy phase
Drug: paclitaxel — Investigator choice of weekly or Q3W during chemotherapy phase
Drug: Avelumab — Given Q3W in combination with carboplatin/paclitaxel during chemotherapy portion
  Arms: Arm C
Drug: Avelumab — Given as single agent in maintenance portion Q2W
  Arms: Arm B; Arm C

SUMMARY:
This is a Phase 3, open-label, international, multi-center, efficacy, and safety study of avelumab in combination with and/or following platinum-based chemotherapy. Eligible patients must have previously untreated, histologically confirmed Stage III-IV epithelial ovarian (EOC), fallopian tube cancer (FTC), or primary peritoneal cancer (PPC) and be candidates for platinum-based chemotherapy.

The primary purpose of the study is to demonstrate if avelumab given as single agent in the maintenance setting following frontline chemotherapy or in combination with carboplatin/paclitaxel is superior to platinum-based chemotherapy alone followed by observation in this population of newly diagnosed ovarian cancer patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed Stage III-IV epithelial ovarian, fallopian tube, or primary peritoneal cancer, including malignant mixed Müllerian tumors with high grade serous component
* Patients must be candidates for platinum based chemotherapy and previously untreated
* Patients must have completed a surgical debulking procedure, or be candidates for neoadjuvant chemotherapy
* Availability of an archival formalin fixed, paraffin embedded (FFPE) tumor tissue block or a minimum of 15 slides
* ECOG PS 0-1
* Adequate hematological, renal, and liver function

Key Exclusion Criteria:

* Non epithelial tumors or ovarian tumors with low malignant potential (ie, borderline tumors) or mucinous tumors
* Prior systemic anti-cancer treatment for EOC, FTC, or PPC including prior immunotherapy with IL 2, IFN α, or anti PD 1, anti PD L1, anti PD L2, anti CD137, or anti cytotoxic T lymphocyte associated antigen 4 (anti CTLA 4) antibody (including ipilimumab), or any other antibody or drug specifically targeting T cell co stimulation or immune checkpoint pathways
* Patients for whom, in the opinion of the Investigator, there is clinical benefit to administer bevacizumab as a first-line treatment and for whom bevacizumab is approved and available in this setting.
* Cancer for which intraperitoneal cytotoxic chemotherapy is planned
* Active autoimmune disease (some exceptions include diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroidism not requiring immunosuppressive treatment)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 998 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2019-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Bradley Monk, MD, Study Chair — Department of Obstetrics and Gynecology University of Arizona Cancer Center, USA; Jonathan Ledermann, MD, Study Chair — UCL Cancer Institute, UK
Locations (304):
- United States (132):
  - Alabama Oncology, Alabaster, Alabama
  - Alabama Oncology, Bessemer, Alabama
  - Alabama Oncology, Bruno Cancer Center, Birmingham, Alabama
  - Alabama Oncology, Birmingham, Alabama
  - Arizona Oncology Associates, PC - HAL, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HAL, Scottsdale, Arizona
  - Arizona Oncology Associates, PC - HAL, Tempe, Arizona
  - Arizona Oncology Associates, PC-HOPE, Tucson, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Oso HomeCare, Irvine, California
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Medical Center, Cedars-Sinai, Los Angeles, California
  - Gynecologic Oncology Associates, Newport Beach, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Hematology-Oncology Medical Group of Orange County, Orange, California
  - Medical Oncology Care Associates, Orange, California
  - St. Joseph Hospital of Orange, Orange, California
  - The Center for Cancer Prevention and Treatment at St. Joseph Hospital of Orange, Orange, California
  - UC Irvine Health, Orange, California
  - University of California, Irvine/UC Irvine Health, Orange, California
  - California Pacific Medical Center - Medical Office Building, San Francisco, California
  - California Pacific Medical Center - Van Ness Campus, San Francisco, California
  - California Pacific Medical Center - Davies Campus, San Francisco, California
  - Bryan Hemming Cancer Care Center - California Pacific Medical Center, San Francisco, California
  - California Pacific Medical Center - Pacific Heights Outpatient Pharmacy, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - California Pacific Medical Center-Research Institute, San Francisco, California
  - Palo Alto Medical Foundation Group, San Francisco, California
  - Sansum Clinic, Santa Barbara, California
  - Sansum Clinic, Solvang, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - C/O Thomas Ferencz, RPh, BCOP, Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Johns Hopkins Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - UHEALTH Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Hospital and Clinics, Miami, Florida
  - Orlando Health Gynecological Cancer Center, Orlando, Florida
  - Orlando Health UF Health Cancer Center, Orlando, Florida
  - Orlando Health, Inc., Orlando, Florida
  - Orlando Health, Inc, Orlando, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Investigational Drug Service, Emory University Clinic, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins University, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Rcca Md Llc, Bethesda, Maryland
  - Rcca Md Llc, Germantown, Maryland
  - SKCCC at Johns Hopkins, Green Spring Station, Lutherville, Maryland
  - Women's Health Specialists of Montgomery County, Rockville, Maryland
  - Holy Cross Resource Center, Silver Spring, Maryland
  - Maryland Oncology Hematology, Silver Spring, Maryland
  - Holy Cross Hospital, Pharmacy, Silver Spring, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Maryland Oncology Hematology, Wheaton, Maryland
  - Massachusetts General Hospital Attn: Svetlana Rashkova, RPh, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center Attn: Nisha Sharma, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute Attn: Vasilika Koci, PharmD, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mercy Ministry Office, Chesterfield, Missouri
  - Mercy - Women's Oncology, Springfield, Missouri
  - Mercy Clinic Cancer and Hematology - Chub O'Reilly Cancer Center, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Summit Medical Group PA, Florham Park, New Jersey
  - University Hospital, Investigational Drug Pharmacy, Newark, New Jersey
  - University Hospital, Newark, New Jersey
  - University Hospital, Ambulatory Care Center, Newark, New Jersey
  - University Hospital, The Cancer Center, Newark, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Medical Arts Radiology, Huntington, New York
  - ProHealth Radiology, Huntington, New York
  - NYU Winthrop Hospital, Clinical Trials Center, Mineola, New York
  - NYU Winthrop Hospital, Gynecologic Oncology, Mineola, New York
  - NYU Winthrop Hospital, Infusion Center, Mineola, New York
  - NYU Winthrop Hospital, Research Pharmacy, Mineola, New York
  - NYU Winthrop Radiology, Mineola, New York
  - Montefiore - Einstein Center for Cancer Care, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Montefiore Medical Center, Centennial Women's Center, The Bronx, New York
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - OSU Wexner Medical Center, Arthur G. James Cancer Hospital & Solove Research Institute, Columbus, Ohio
  - OSU Wexner Medical Center, Investigational Drug Services, Columbus, Ohio
  - OSU Wexner Medical Center, Stefanie Spielman Comprehensive Breast Center, Columbus, Ohio
  - Oncology Hematology Care, Inc., Fairfield, Ohio
  - OSU Wexner Medical Center, Gynecologic Oncology at Mill Run, Hilliard, Ohio
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Asante Three Rivers Medical Center, Grants Pass, Oregon
  - Hematology Oncology Associates, Grants Pass, Oregon
  - Asante Pharmacy, Medford, Oregon
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Hematology Oncology Associates, Medford, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Magee-Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute Investigational Drug Service, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Tennessee Oncology, PLLC, Dickson, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Shelbyville, Tennessee
  - Tennessee Oncology, PLLC, Smyrna, Tennessee
  - Texas Oncology-Austin Central, Austin, Texas
  - Texas Oncology - South Austin, Austin, Texas
  - Texas Oncology Bedford, Bedford, Texas
  - Parkland Health and Hospital System, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - UT Southwestern Medical Center-Clements University Hospital, Dallas, Texas
  - UT Southwestern Medical Center-Zale Lipshy University Hospital, Dallas, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - US Oncology Investigational Products Center (IPC), Irving, Texas
  - US Oncology Investigational Products Center, Irving, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - Utah Cancer Specialists, Layton, Utah
  - Utah Cancer Specialists, Murray, Utah
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Utah Cancer Specialists, West Jordan, Utah
  - Emily Couric Cancer Center, Charlottesville, Virginia
- Bulgaria (2):
  - MHAT for Female Health-Nadezhda OOD, Sofia
  - Shato Ead, Sofia
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre-Glen Site, Montreal, Quebec
  - Oncology Pharmacy McGill University Health Centre, Montreal, Quebec
  - CHU de Quebec-Universite Laval, Québec, Quebec
- Croatia (2):
  - Klinicki bolnicki centar Split, Split
  - Klinicki bolnicki centar Sestre milosrdnice, Zagreb
- Estonia (5):
  - East Tallinn Central Hospital, Tallinn
  - East-Tallinn Central Hospital, Center of Oncology, Tallinn
  - North Estonia Medical Centre Foundation, Pharmacy, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Hematology and Oncology Clinic, Tartu
- Germany (11):
  - Zentralapotheke Zytostatika, Chemnitz
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Radiologie Uniklinik Koeln, Cologne
  - Uniklinik Koeln Apotheke, Cologne
  - Uniklinik Koeln Klinik fuer Frauenheilkunde und Geburtshilfe, Cologne
  - Johannes Apotheke Klinikversorgung, Gröbenzell
  - Radiologie Muenchen, München
  - Frauenklinik am Rotkreuzklinikum Muenchen, München
  - Diagnostische und Interventionelle Radiologie, Potsdam
  - Klinikum Ernst von Bergmann gGmbH, Potsdam
  - Universitaetsklinikum Wuerzburg Frauenklinik und Poliklinik, Würzburg
- Hong Kong (2):
  - Queen Elizabeth Hospital, Hong Kong
  - The University of Hong Kong, Hong Kong
- Hungary (4):
  - Semmelweis Egyetem Onkologiai Kozpont, Budapest
  - Debreceni Egyetem Klinikai Gyogyszertar, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Szuleszeti es Nogyogyaszati Klinika, Debrecen
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Onkologiai Kozpont, Szolnok
- Ireland (8):
  - Mater Misericordiae University Hospital, Dublin, Dublin
  - Mater Private Hospital, Dublin, Dublin
  - Bon Secours Hospital Ireland, Cork
  - Bon Secours Hospital, Cork
  - Pharmacy Department, St James's Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - St James's Hospital, Dublin
- Italy (9):
  - Azienda Ospedaliero -Universitaria di Bologna Policlinico S. Orsola - Malpighi, Bologna, BO
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola - Malpighi, Bologna, BO
  - E.O. Ospedali Galliera, Genova, GE
  - Farmacia Galliera, Genova, GE
  - Istituto Europeo di Oncologia, Milan, MI
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - Azienda Socio Sanitaria Territoriale ASST della Valtellina e dell Alto Lario, Sondrio, SO
  - Istituto Nazionale Tumori Napoli IRCCS Fondazione Pascale, Napoli
  - Dip.to per la Tutela della Salute della Donna, della Vita Nascente, del Bambino e dell'Adolescente, Roma
- Japan (16):
  - The Jikei University Kashiwa Hospital, Kashiwa-shi, Chiba
  - Shikoku Cancer Center, Matsuyama, Ehime
  - Ehime University Hospital, Tōon, Ehime
  - Kurume University Hospital, Kurume, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Tokai University Hospital, Isehara, Kanagawa
  - Kyoto University Hospital, Sakyo-ku, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - National Defense Medical College Hospital, Tokorozawa, Saitama
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Jikei University Hospital, Minato-ku, Tokyo
  - Niigata Cancer Center Hospital, Niigata
- Latvia (7):
  - Daugavpils Regional Hospital, Oncology Department (11 floor), Daugavpils
  - Daugavpils Regional Hospital, Daugavpils
  - Natalja Goncarova -Radiology Services, Daugavpils
  - Inga Vigule-Radiology services, Liepāja
  - Liepaja Regional hospital, Liepāja
  - Pauls Stradins Clinical University Hospital, Riga
  - Medical Society "ARS" Ltd, Riga
- Mexico (2):
  - Instituto Nacional de Cancerologia, Mexico City, Mexico City
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
- Netherlands (7):
  - Academisch Medisch Centrum, Amsterdam
  - Pharmacy Universitair Medisch Centrum Groningen, Groningen
  - Universitair Medisch Centrum Groningen, Groningen
  - LUMC, Leiden
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Pharmacy Zuyderland Medisch Centrum, Sittard-Geleen
  - Zuyderland Medisch Centrum, Sittard-Geleen
- Poland (8):
  - Szpitale Pomorskie Sp. z.o.o., Apteka Szpitalna, Gdynia
  - Szpitale Pomorskie, Sp. z o. o., Oddzial Onkologii i Radioterapii, Gdynia
  - Centrum Onkologii, Instytut im. M. Sklodowskiej-Curie, Oddzial w Krakowie, Apteka Szpitalna, Krakow
  - Centrum Onkologii, Instytut im.M.Sklodowskiej-Curie, Oddzial w Krakowie, Krakow
  - Wojewodzki Szpital Specjalistyczny w Olsztynie. Apteka Szpitalna, Olsztyn
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Opolskie Centrum Onkologii im. prof. Tadeusza Koszarowskiego w Opolu, Opole
  - Ginekologiczno - Polozniczy Szpital Kliniczny Uniwersytetu Medycznego im. Karola Marcinkowskiego w, Poznan
- Romania (3):
  - SC Medisprof SRL, Cluj-Napoca, Cluj
  - SC Oncolab SRL, Craiova, Dolj
  - SC Centrul de Oncologie Euroclinic SRL, Iași
- Russia (11):
  - Limited liability company (LLC) EVIMED, Chelyabinsk, Chelyabinsk Oblast
  - State Budgetary Healthcare Institution, Chelyabinsk, Chelyabinsk Oblast
  - Regional Budgetary Healthcare Institution (RBHI) Ivanovo Regional Oncology Dispensary, Ivanovo, Ivanovo Oblast
  - FSBI - NMRRC Minzdrav Russia at the branch A.F.Tsyb Medical Radiological Research Centre, Obninsk, Kaluga Oblast
  - SBHI Orenburg Regional Clinical Oncology Dispensary (SBHI ORCOD), Orenburg, Orenburg Oblast
  - SAHI "Republican Clinical Oncology Dispensary of the MoH of TR", Kazan', Tatarstan Republic
  - SBHI Moscow Clinical Scientific and Practical Centre of Moscow City Healthcare Department, Moscow
  - FSBI National Research Medical Center of Oncology N.A., Moscow
  - Clinic, Moscow
  - Limited liability company VitaMed-LLC VitaMed, Moscow
  - SBHI Saint-Petersburg Clinical Scientific - Practice Center of Specialized Types of Medical Care, Saint Petersburg
- Singapore (3):
  - National University Hospital, Singapore
  - National University Hospital, Pharmacy @ NCIS, Singapore
  - Raffles Hospital, Singapore
- Slovakia (5):
  - NsP sv. Jakuba, n.o. , Bardejov, Bardejov
  - Onkologicky ustav sv. Alzbety a.s., Bratislava
  - Narodny onkologicky ustav, Bratislava
  - Vychodoslovensky onkologicky ustav, a.s., Košice
  - POKO Poprad s.r.o., Poprad
- South Korea (15):
  - Center for Uterine Cancer, National Cancer Center, Goyang-si, Gyeonggi-do
  - Clinical Trial Pharmacy, National Cancer Center, Goyang-si, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Clinical Trial Pharmacy, Seongnam-si, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Korea University Anam Hospital, Clinical Trial Pharmacy, Seoul
  - Korea University Anam Hospital, Seoul
  - CTC Cancer Pharmacy, Seoul National University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Clinical Research Pharmacy, Seoul
  - Asan Medical Center, Seoul
  - Clinical Trial Pharmacy, Samsung Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Clinical Trial Pharmacy, Korea University Guro Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Switzerland (4):
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - Oncology Institute of Southern Switzerland (IOSI), Bellinzona, Canton Ticino
  - Ospedale San Giovanni, Bellinzona, Canton Ticino
  - Radiologia ORBV, Bellinzona, Canton Ticino
- Taiwan (11):
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Clinical Trial Pharmacy, MacKay Memorial Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Clinical Trial Pharmacy, Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Clinical Trial Pharmacy, Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan
  - Chemotherapy Pharmacy, Chang Gung Memorial Hospital - Linkou Branch, Taoyuan
- Turkey (Türkiye) (6):
  - Baskent University Adana Training and Research Hospital, Adana
  - Baskent University Ankara Hospital, Department of Oncology, Ankara
  - Bezmialem Vakif University Medical Faculty Hospital, Istanbul
  - Istanbul University Oncology Institute, Istanbul
  - Istanbul University Cerrahpasa-Cerrahpasa Medical Faculty, Istanbul
  - Ege University Faculty of Medicine Hospital, Izmir
- Ukraine (6):
  - Communal Institution Chernivtsi Regional Clinical Oncology Dispensary, Chernivtsi
  - Cl Dnipropetrovsk City Multifield Clinical Hospital, Dnipropetrovsk
  - Municipal Institution Kryviy Rih Oncology Center of Dnipropetrovsk regional Council, Kryviy Rig
  - Clinic of National Cancer Institute, Kyiv
  - CNE of Lviv Regional Council "Lviv Oncological Regional Therapeutical and Diagnostic Centre", Lviv
  - Central Municipal Clinical Hospital, Municipal oncology center, therapeutics department, Uzhhorod
- United Kingdom (19):
  - Torbay and South Devon NHS Foundation Trust, Torquay, Devon
  - East Kent Hospitals University NHS Foundation Trust, Margate, KENT
  - University College London Hospital NHS Foundation Trust, Islington, London
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral, Merseyside
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral, Merseyside
  - East and North Hertfordshire NHS Trust, Northwood, Middlesex
  - Oxford University Hospitals NHS Foundation Trust, Headington, Oxford
  - Royal Surrey County Hospital NHS Foundation Trust, Guildford, Surrey
  - Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - University Hospitals Bristol NHS Foundation trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - University College London Hospital NHS Foundation Trust, London
  - Guy's & St Thomas' NHS Foundation Trust, London
  - Royal Marsden NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - University College London Hospital, London
  - The Christie Hospital NHS Foundation Trust, Manchester
  - Baxter Healthcare, Stockport

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Monk BJ, Colombo N, Oza AM, Fujiwara K, Birrer MJ, Randall L, Poddubskaya EV, Scambia G, Shparyk YV, Lim MC, Bhoola SM, Sohn J, Yonemori K, Stewart RA, Zhang X, Perkins Smith J, Linn C, Ledermann JA. Chemotherapy with or without avelumab followed by avelumab maintenance versus chemotherapy alone in patients with previously untreated epithelial ovarian cancer (JAVELIN Ovarian 100): an open-label, randomised, phase 3 trial. Lancet Oncol. 2021 Sep;22(9):1275-1289. doi: 10.1016/S1470-2045(21)00342-9. Epub 2021 Aug 4. PMID 34363762
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991010

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy Followed by Avelumab: In chemotherapy phase (CP),based on investigator's decision,participants received either:paclitaxel 175 milligrams per square meter (mg/m2) intravenous (IV) infusion,followed by carboplatin dose at area under curve (AUC) 5 or 6,IV infusion (carboplatin dose (mg) = Target AUC (mg*min/mL) x (glomerular filtration rate[GFR] mL/min + 25),and maximum carboplatin dose = target AUC x (150 mL/min) on Day 1 of Cycles 1 to 6; or Paclitaxel 80 mg/m2 IV infusion over 1 hour on Days 1, 8, and 15, along with carboplatin dose at AUC 5 or 6, IV infusion over 1 hour on Day 1 of Cycle 1 to 6 (1 cycle=21 days). After completion of CP, participants without evidence of disease progression, received avelumab 10 mg/kg, over 1 hour IV infusion,once every 2 weeks on Days 1, 15, and 29 (1 cycle=42 days) in maintenance phase (MP) until confirmed progressive disease,unacceptable toxicity, or withdrawal of consent, or a maximum duration of 24 months. Participants were then followed up to a maximum of 36 months.
- Chemotherapy + Avelumab Followed by Avelumab: In CP, based on investigator's decision, participants received either:paclitaxel 175 mg/m2,IV,followed by carboplatin dose at AUC 5 or 6,IV (carboplatin dose [milligrams](mg) = Target AUC (mg*min/mL) x GFR mL/min + 25),and maximum carboplatin dose = target AUC x (150 mL/min) on Day 1 of Cycles 1 to 6;or Paclitaxel 80 mg/m2 IV infusion over 1 hour on Days 1, 8, and 15, along with carboplatin dose at AUC 5 or 6, IV infusion over 1 hour on Day 1 of Cycle 1 to 6 along with Avelumab 10 mg/kg administered as a 1-hour IV infusion once every 3 weeks for Cycle 1 to 6 ( 1 cycle=21 days).After completion of CP, participants without evidence of disease progression, received Avelumab IV, 10 mg/kg, once every 2 weeks on Days 1, 15, and 29 ( 1 cycle=42 days) in MP until confirmed progressive disease (PD), unacceptable toxicity, or withdrawal of consent, or a maximum duration of 24 months. Participants were then followed up to a maximum of 36 months.
- Chemotherapy Followed by Observation: In CP, based on investigator's decision, participants received either: paclitaxel 175 mg/m2, IV infusion, followed by carboplatin dose at AUC 5 or 6, IV infusion (carboplatin dose [milligrams](mg) = Target AUC [milligrams*minute per milliliter] (mg*min/mL) x GFR mL/min + 25), and maximum carboplatin dose = target AUC x (150 mL/min) on Day 1 of Cycles 1 to 6; or Paclitaxel 80 mg/m2 IV infusion over 1 hour on Days 1, 8, and 15, along with carboplatin dose at AUC 5 or 6, IV infusion over 1 hour on Day 1 of Cycle 1 to 6. Each cycle was of 21 days (3 weeks). After completion of CP, participants were followed for survival status until death or until study completion, whichever was earlier or a maximum duration of 24 months in observation phase. Participants were then followed up to a maximum of 36 months.
Period: Chemotherapy Phase (CP)
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Started | 332 | 331 | 335
Safety Population (Participants who had received at least one dose of study drug) | 328 | 329 | 334
Completed | 280 | 294 | 289
Not Completed | 52 | 37 | 46
Not completed — Adverse Event | 9 | 14 | 13
Not completed — Death leading to discontinuation | 5 | 4 | 1
Not completed — Global deterioration of health status | 3 | 2 | 1
Not completed — No longer met eligibility criteria | 4 | 2 | 1
Not completed — Physician's decision | 5 | 0 | 4
Not completed — Progressive disease | 11 | 7 | 10
Not completed — Withdrawal by Subject | 13 | 8 | 15
Not completed — Other | 2 | 0 | 1
Period: Maintenance Phase (MP)
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Started | 267 (Included participants without evidence of disease progression at the end of Chemotherapy phase.) | 288 (Included participants without evidence of disease progression at the end of Chemotherapy phase.) | 0 (After completing CP, participants moved to observation phase. MP was not applicable for this arm.)
Completed | 1 | 1 | 0
Not Completed | 266 | 287 | 0
Not completed — Adverse Event | 21 | 26 | 0
Not completed — Death leading to discontinuation | 1 | 1 | 0
Not completed — Global deterioration of health status | 5 | 3 | 0
Not completed — No longer met eligibility criteria | 0 | 1 | 0
Not completed — Physician's decision | 6 | 7 | 0
Not completed — Progressive disease | 100 | 88 | 0
Not completed — Other | 2 | 1 | 0
Not completed — Withdrawal by Subject | 17 | 20 | 0
Not completed — Study terminated by sponsor | 114 | 140 | 0
Period: Observation Phase (OP)
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Started | 0 (After completing MP, participants moved to follow-up phase. OP was not applicable.) | 0 (After completing MP, participants moved to follow-up phase. OP was not applicable.) | 284 (Included participants without evidence of disease progression at the end of Chemotherapy phase.)
Completed | 0 | 0 | 2
Not Completed | 0 | 0 | 282
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Death leading to discontinuation | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 9
Not completed — Progressive disease | 0 | 0 | 92
Not completed — Study terminated by sponsor | 0 | 0 | 135
Not completed — Withdrawal by Subject | 0 | 0 | 34
Not completed — Global deterioration of health status | 0 | 0 | 1
Not completed — Other | 0 | 0 | 7
Period: Follow-up Phase
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Started | 238 (Participants not completing MP could also start this phase.) | 263 (Participants not completing MP could also start this phase.) | 39 (Participants not completing OP could also start this phase.)
Completed | 103 | 91 | 20
Not Completed | 135 | 172 | 19
Not completed — Adverse Event | 3 | 1 | 1
Not completed — Other | 4 | 6 | 4
Not completed — Withdrawal by Subject | 19 | 17 | 5
Not completed — Study terminated by sponsor | 100 | 138 | 6
Not completed — Lost to Follow-up | 2 | 3 | 0
Not completed — Death leading to discontinuation | 7 | 7 | 3
Period: Long-term Follow-up Phase
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Started | 139 (Participants not completing follow-up phase could also start this phase.) | 112 (Participants not completing follow-up phase could also start this phase.) | 135 (Participants not completing follow-up could also start this phase.)
Completed | 0 | 0 | 0
Not Completed | 139 | 112 | 135
Not completed — Death leading to discontinuation | 20 | 17 | 11
Not completed — Lost to Follow-up | 8 | 4 | 3
Not completed — Study terminated by sponsor | 105 | 80 | 112
Not completed — Withdrawal by Subject | 6 | 9 | 9
Not completed — Other | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation | Total
Number analyzed (Participants) | 332 | 331 | 335 | 998
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean | 58.34 (11.00) | 58.16 (10.85) | 57.10 (11.27) | 57.86 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 332 | 331 | 335 | 998
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 4 | 1 | 7
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 86 | 82 | 95 | 263
  White | 236 | 238 | 236 | 710
  Other | 7 | 7 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Assessed by Blinded Independent Central Review (BICR)
Description: BICR assessed PFS: Duration from randomization until disease progression or death. PFS data was censored on the date of the last adequate tumor assessment for participants who did not have an event (progression of disease or death), who started a new anti-cancer therapy prior to an event or for participants with an event after 2 or more missing tumor assessments. Progression as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1: as at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 millimeters (mm). The appearance of one or more new lesions was also considered progression. Analysis was performed using Kaplan-Meier method.
Time Frame: Baseline to progression of disease or discontinuation from the study or death, whichever occurred first (maximum duration of 27 months)
Population: The full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 332 | 331 | 335
months | 16.8 [13.5 to NA] — The upper limit of 95% CI was not estimable due to limited number of events. | 18.1 [14.8 to NA] — The upper limit of 95% CI was not estimable due to limited number of events. | NA [18.2 to NA] — The median and upper limit of 95% CI was not estimable due to limited number of events.
Statistical Analysis 1: Comparison: Chemotherapy Followed by Avelumab vs Chemotherapy Followed by Observation; Test type: Superiority; p = 0.9890, Log Rank — One-sided log-rank test was used; Analysis was performed using a Cox's Proportional Hazard model stratified by the randomization strata and a stratified log-rank test; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [1.051 to 1.946]
Statistical Analysis 2: Comparison: Chemotherapy + Avelumab Followed by Avelumab vs Chemotherapy Followed by Observation; Test type: Superiority; p = 0.7935, Log Rank — One-sided log-rank test was used; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.832 to 1.565]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time (in months) from the date of randomization to the date of death due to any cause. Participants last known to be alive were censored at date of last contact. Analysis was performed using Kaplan-Meier method.
Time Frame: Baseline to discontinuation from the study or death, whichever occurred first (maximum duration of 27 months)
Population: The full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 332 | 331 | 335
months | NA [NA to NA] — Median and 95% CI were not estimable due to limited number of events. | NA [NA to NA] — Median and 95% CI were not estimable due to limited number of events. | NA [NA to NA] — Median and 95% CI were not estimable due to limited number of events.
Statistical Analysis 1: Comparison: Chemotherapy Followed by Avelumab vs Chemotherapy Followed by Observation; Test type: Superiority; p = 0.8848, Log Rank — One-sided log-rank test was used; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.53, 95% CI 2-sided [0.760 to 3.080]
Statistical Analysis 2: Comparison: Chemotherapy + Avelumab Followed by Avelumab vs Chemotherapy Followed by Observation; Test type: Superiority; p = 0.8953, Log Rank — One-sided log-rank test was used; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.55, 95% CI 2-sided [0.776 to 3.111]

3. Secondary Outcome: Progression-Free Survival (PFS) as Assessed by Investigator
Description: Investigator assessed PFS was defined as time (in months) from date of randomization to the first documentation of disease progression or death (due to any cause), whichever occurred first. Progression as per RECIST 1.1, was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression. Analysis was performed using a Cox's Proportional Hazard model stratified by the randomization strata and a stratified log-rank test.
Time Frame: as for outcome 1
Population: The full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 332 | 331 | 335
months | 13.8 [12.1 to 15.9] | 16.1 [13.9 to 19.4] | 15.0 [13.2 to 18.7]
Statistical Analysis 1: Comparison: Chemotherapy Followed by Avelumab vs Chemotherapy Followed by Observation; Test type: Other; p = 0.9278, Log Rank — One-sided log-rank test was used; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.935 to 1.578]
Statistical Analysis 2: Comparison: Chemotherapy + Avelumab Followed by Avelumab vs Chemotherapy Followed by Observation; Test type: Other; p = 0.2367, Log Rank — One-sided log-rank test was used; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.688 to 1.189]

4. Secondary Outcome: Percentage of Participants With Objective Response as Assessed by Investigator
Description: Investigator assessed objective response according to RECIST version 1.1, was defined as participants with confirmed best overall response of complete response (CR) or partial response (PR). CR was defined as disappearance of all target and non-target lesions, and sustained for at least 4 weeks. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 mm. PR was defined as at least 30% decrease in the sum of the longest dimensions of target lesions taking as reference the baseline sum longest dimensions.
Time Frame: Baseline to progression of disease, start of new anti-cancer therapy or discontinuation from study or death, whichever occurred first (maximum duration of 27 months)
Population: The full analysis set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 332 | 331 | 335
percentage of participants | 25.9 [21.3 to 31.0] | 31.1 [26.2 to 36.4] | 27.8 [23.0 to 32.9]

5. Secondary Outcome: Percentage of Participants With Objective Response as Assessed by Blinded Independent Central Review (BICR)
Description: BICR assessed objective response according to RECIST version 1.1, was defined as participants with confirmed best overall response of CR or PR. CR was defined as disappearance of all target and non-target lesions, and sustained for at least 4 weeks. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least 30% decrease in the sum of the longest dimensions of target lesions taking as reference the baseline sum longest dimensions.
Time Frame: as for outcome 4
Population: The full analysis set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 332 | 331 | 335
percentage of participants | 30.4 [25.5 to 35.7] | 36.0 [30.8 to 41.4] | 30.4 [25.6 to 35.7]

6. Secondary Outcome: Duration of Response (DOR) as Assessed by Investigator
Description: Investigator assessed DOR: time (in months) from the first documentation of objective response (confirmed CR or PR) to the date of first documentation of PD or death due to any cause. As per RECIST version 1.1, CR was defined as disappearance of all target and non-target lesions, and sustained for at least 4 weeks. Any pathological lymph nodes (target or non-target) must have reduction in short axis to <10 mm. PR: at least 30% decrease in the sum of the longest dimensions of target lesions taking as reference the baseline sum longest dimensions. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression. Analysis was performed using Kaplan-Meier method.
Time Frame: First response subsequently confirmed to progression of disease or start of new anti-cancer therapy or discontinuation from the study or death, whichever occurred first (maximum duration of 27 months)
Population: Analysis was performed on subset of randomized participants, who had objective response, as assessed by Investigator.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 86 | 103 | 93
months | 10.6 [8.3 to 20.2] | NA [11.7 to NA] — Median and upper limit of 95% CI was not estimable due to limited number of events. | 15.4 [8.3 to 18.4]

7. Secondary Outcome: Duration of Response (DOR) as Assessed by Blinded Independent Central Review (BICR)
Description: BICR assessed DOR: time (in months) from the first documentation of objective response (confirmed CR or PR) to the date of first documentation of PD or death due to any cause. As per RECIST version 1.1, CR was defined as disappearance of all target and non-target lesions, and sustained for at least 4 weeks. Any pathological lymph nodes (target or non-target) must have reduction in short axis to <10 mm. PR: at least 30% decrease in the sum of the longest dimensions of target lesions taking as reference the baseline sum longest dimensions. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression. Analysis was performed using Kaplan-Meier method.
Time Frame: as for outcome 6
Population: Analysis was performed on subset of randomized participants, who had objective response, as assessed by BICR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 101 | 119 | 102
months | 11.9 [8.9 to NA] — The upper limit of 95% CI was not estimable due to limited number of events. | 14.5 [11.7 to NA] — The upper limit of 95% CI was not estimable due to limited number of events. | NA [16.1 to NA] — The median and upper limit of 95% CI was not estimable due to limited number of events.

8. Secondary Outcome: Maintenance Progression-Free Survival as Assessed by Blinded Independent Central Review (BICR)
Description: BICR assessed maintenance PFS was defined as the time from Cycle 1 Day 1 of the maintenance phase to the date of the first documentation of PD or death due to any cause, whichever occurs first. It was defined, for participants who proceeded to maintenance phase and who did not have disease progression by BICR during the chemotherapy phase. As per RECIST version 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression. Analysis was performed using Kaplan-Meier method.
Time Frame: From Day 1 of Cycle 1 (42 days) of maintenance phase to progression of disease or death, whichever occurred first (maximum duration of 27 months)
Population: The analysis set included randomized participants who proceeded to maintenance phase and who did not have PD by BICR assessment during the chemotherapy phase.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 248 | 267 | 247
months | 13.6 [9.3 to NA] — The upper limit of 95% CI was not estimable due to limited number of events. | 13.8 [11.1 to NA] — The upper limit of 95% CI was not estimable due to limited number of events. | NA [13.8 to NA] — The median and upper limit of 95% CI was not estimable due to limited number of events.

9. Secondary Outcome: Maintenance Progression-Free Survival (PFS) as Assessed by Investigator
Description: Investigator assessed maintenance PFS was defined as the time from Cycle 1 Day 1 of the maintenance phase to the date of the first documentation of PD or death due to any cause, whichever occurs first. It was defined, for participants who proceeded to maintenance phase and who did not have disease progression by investigator during the chemotherapy phase. As per RECIST version 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression. Analysis was performed using Kaplan-Meier method
Time Frame: as for outcome 8
Population: The analysis set included randomized participants who proceeded to maintenance phase and who did not have PD by investigator assessment during the chemotherapy phase.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 252 | 271 | 252
months | 10.4 [8.2 to 13.6] | 11.6 [9.9 to 13.8] | 12.7 [9.5 to NA] — The upper limit of 95% CI was not estimable due to limited number of events.

10. Secondary Outcome: Percentage of Participants With Pathological Complete Response (pCR)
Description: pCR was defined (for neoadjuvant participants who underwent interval debulking surgery [IDS]), as the chemotherapy response score 3 (CSR3), based on a study by Bohm et al, 2015. CSR3 was defined as complete or near-complete response with no residual tumor or minimal irregularly scattered tumor foci seen as individual cells, cell groups, or nodules up to 2 mm. Complete or near-complete response was defined as complete or near-complete microscopic disappearance of invasive tumor/ residual disease.
Time Frame: as for outcome 1
Population: Analysis was performed on a subset of randomized participants which included neoadjuvant participants who underwent IDS.
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 108 | 115 | 116
percentage of participants | 15.7 | 17.4 | 25.9

11. Secondary Outcome: Progression-Free Survival 2 (PFS2)
Description: PFS2 was defined as time (in months) from the date of randomization to the start of second subsequent treatment after first documentation of PD, or death from any cause, whichever occurred first. Progression as per RECIST version 1.1, was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression. Analysis was performed using Kaplan-Meier method.
Time Frame: Baseline up to start of second subsequent treatment after first PD or discontinuation from study or death, which ever occured first (maximum duration of 27 months)
Population: The trial was terminated due to crossing of futility boundaries for both experimental arms as compared to the control arm at the pre-specified interim analysis for PFS based on BICR assessment. Subsequently, the data for this outcome measure was not collected and analyzed.
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Progression-Free Survival (PFS) as Assessed by Gynecological Cancer Intergroup (GCIG) Criteria
Description: PFS by GCIG was assessed by both RECIST 1.1 and cancer antigen 125 (CA-125). It was defined as time from randomization to first documentation of disease progression (PD) or death, whichever occurred first. As per RECIST 1.1, PD: greater than or equal to (>=) 20 % increase in the sum of diameters of target lesions, taking as reference the smallest sum on study with absolute increase >= 5 millimeters. PD based on serum CA-125 was defined as (i) participants with elevated CA-125 pretreatment and normalization of CA-125, (ii) participants with CA-125 in the reference range before treatment; (i) and (ii) must have showed CA-125 >= 2 times the upper limit of the reference range on 2 occasions >= 1 week apart, or (iii) participants with elevated CA-125 before treatment, which never normalized, showed CA-125 >= 2 times the nadir value on 2 occasions >= 1 week apart. Censoring date for PFS by GCIG was the latest of the censoring dates for PFS by RECIST 1.1 and PFS by CA-125.
Time Frame: Baseline until disease progression by GCIG criteria or start of new anti-cancer therapy or discontinuation from the study or death, whichever occurred first (maximum duration of 27 months)
Population: as for outcome 11
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) Graded Based on, National Cancer Institute Common Terminology Criteria (NCI-CTCAE), Version 4.03
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per NCI-CTCAE version 4.03, Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE. Treatment-emergent events are events between first dose of study drug and up to 36 months that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline to discontinuation from the study or death, whichever occurred first (maximum duration of 36 months)
Population: The safety analysis set included all participants who had received at least one dose of study drug. Here "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 323 | 328 | 321
Participants
  Grade 1 | 11 | 13 | 15
  Grade 2 | 89 | 77 | 96
  Grade 3 | 151 | 148 | 131
  Grade 4 | 67 | 84 | 76
  Grade 5 | 5 | 6 | 3

14. Secondary Outcome: Number of Participants With Laboratory Abnormalities Greater Than or Equal to (>=) Grade 3, Based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE), Version 4.03
Description: As per NCI-CTCAE v 4.03, Grade 3 and above criteria were; Hematology [Anemia - Grade 3: hemoglobin <8.0 grams per deciliter (g/dL), <4.9 millimoles per liter (mmol/L), <80 grams per liter (g/L), transfusion indicated, Grade 4: life-threatening consequences, urgent intervention indicated, Grade 5: death; platelet count decreased- Grade 3:<50.0 to 25.0*10^9/Liters(L), Grade 4: <25.0*10^9/L; lymphocyte count decreased-Grade 3: <0.5-0.2*10^9/L, Grade 4: <0.2*10^9/L; neutrophil count decreased-Grade 3: <1.0 to 0.5*10^9 /L, Grade 4: <0.5*10^9/L]. Chemistry [creatinine increased-Grade 3: >3.0 to 6.0*upper limit of normal (ULN), Grade 4: >6.0*ULN; serum amylase increased, lipase increased-Grade 3: >2.0 - 5.0*ULN, Grade 4: >5.0*ULN]. Liver function [aspartate aminotransferase (AST) and alanine aminotransferase (ALT)-Grade 3: >5.0 to 20.0*ULN, Grade 4: >20.0*ULN].
Time Frame: Baseline to discontinuation from the study or death, whichever occurred first (maximum duration of 27 months)
Population: The safety analysis set included all participants who received at least one dose of study drug. Here, 'Number analyzed' = Participants evaluable for this outcome measure for each specified row.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 328 | 329 | 334
Participants
  Anemia: number analyzed (Participants) | 326 | 326 | 328
  Anemia | 73 | 68 | 63
  Platelet Count Decreased: number analyzed (Participants) | 326 | 326 | 328
  Platelet Count Decreased | 20 | 35 | 38
  Lymphocyte Count Decreased: number analyzed (Participants) | 326 | 326 | 328
  Lymphocyte Count Decreased | 35 | 63 | 29
  Neutrophil Count Decreased: number analyzed (Participants) | 326 | 326 | 328
  Neutrophil Count Decreased | 144 | 159 | 156
  Creatinine Increased: number analyzed (Participants) | 324 | 326 | 327
  Creatinine Increased | 2 | 7 | 0
  Serum Amylase Increased: number analyzed (Participants) | 321 | 322 | 326
  Serum Amylase Increased | 5 | 9 | 10
  Lipase Increased: number analyzed (Participants) | 323 | 323 | 325
  Lipase Increased | 19 | 24 | 11
  ALT or AST: number analyzed (Participants) | 324 | 326 | 327
  ALT or AST | 0 | 1 | 0

15. Secondary Outcome: Change From Baseline in Vital Signs - Blood Pressure at Day 1 of Cycles 2, 3, 4 in Chemotherapy Phase; Days 1, 15 and 29 of Cycles 1 and 2 in Maintenance/ Observation Phase and at End of Treatment
Description: Vital signs included blood pressure and pulse rate. Blood pressure included sitting diastolic blood pressure (DBP) and sitting systolic blood pressure (SBP). MP is applicable only for two arms 'Chemotherapy followed by Avelumab' and 'Chemotherapy + Avelumab followed by Avelumab'. OP is applicable only for third arm 'Chemotherapy followed by Observation'. Category titles 'MP/OP' imply which ever phase was applicable for the respective reporting arms.
Time Frame: Baseline, first 3 months of Chemotherapy Phase (CP): Day 1 of Cycles 2, 3 and 4 (each cycle 21 days); Maintenance/Observation Phase (MP/OP): Days 1, 15 and 29 of Cycles 1 and 2 (each cycle 42 days) and at end of treatment (up to 27 months)
Population: The safety analysis set included all participants who had received at least one dose of study drug. Here "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and 'Number analyzed' = participants evaluable for this outcome measure at specified rows.
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 318 | 317 | 316
millimeters of mercury
  CP: Change at Day 1, Cycle 2: Sitting DBP: number analyzed (Participants) | 310 | 305 | 301
  CP: Change at Day 1, Cycle 2: Sitting DBP | 0.00 (9.28) | 0.10 (9.86) | 0.70 (9.33)
  CP: Change at Day 1, Cycle 3: Sitting DBP: number analyzed (Participants) | 305 | 299 | 295
  CP: Change at Day 1, Cycle 3: Sitting DBP | -0.50 (10.18) | 0.50 (10.84) | 1.00 (9.69)
  CP: Change at Day 1, Cycle 4: Sitting DBP: number analyzed (Participants) | 287 | 291 | 289
  CP: Change at Day 1, Cycle 4: Sitting DBP | -0.10 (10.48) | -0.50 (10.89) | -0.40 (10.19)
  MP/OP: Change at Day 1, Cycle 1: Sitting DBP: number analyzed (Participants) | 253 | 266 | 253
  MP/OP: Change at Day 1, Cycle 1: Sitting DBP | -2.20 (10.36) | -1.30 (10.74) | -0.90 (10.54)
  MP/OP: Change at Day 15, Cycle 1: Sitting DBP: number analyzed (Participants) | 241 | 249 | 3
  MP/OP: Change at Day 15, Cycle 1: Sitting DBP | -2.10 (10.04) | -1.80 (10.57) | -9.70 (5.69)
  MP/OP: Change at Day 29, Cycle 1: Sitting DBP: number analyzed (Participants) | 233 | 249 | 3
  MP/OP: Change at Day 29, Cycle 1: Sitting DBP | -1.70 (10.29) | -1.80 (11.24) | -8.30 (6.03)
  MP/OP: Change at Day 1, Cycle 2: Sitting DBP: number analyzed (Participants) | 229 | 247 | 226
  MP/OP: Change at Day 1, Cycle 2: Sitting DBP | -2.30 (10.26) | -1.70 (10.63) | -0.70 (10.67)
  MP/OP: Change at Day 15, Cycle 2: Sitting DBP: number analyzed (Participants) | 219 | 236 | 0
  MP/OP: Change at Day 15, Cycle 2: Sitting DBP | -2.00 (10.71) | -2.40 (10.82) |
  MP/OP: Change at Day 29, Cycle 2: Sitting DBP: number analyzed (Participants) | 215 | 225 | 0
  MP/OP: Change at Day 29, Cycle 2: Sitting DBP | -2.60 (10.86) | -1.90 (10.16) |
  Change at EOT : Sitting DBP: number analyzed (Participants) | 137 | 116 | 120
  Change at EOT : Sitting DBP | -0.70 (11.36) | 0.00 (12.45) | 0.70 (10.00)
  CP: Change at Day 1, Cycle 2: Sitting SBP: number analyzed (Participants) | 310 | 305 | 301
  CP: Change at Day 1, Cycle 2: Sitting SBP | 2.30 (14.91) | 0.70 (15.32) | 1.00 (14.00)
  CP: Change at Day 1, Cycle 3: Sitting SBP: number analyzed (Participants) | 305 | 299 | 295
  CP: Change at Day 1, Cycle 3: Sitting SBP | 1.50 (14.00) | -0.30 (15.48) | 1.70 (14.80)
  CP: Change at Day 1, Cycle 4: Sitting SBP: number analyzed (Participants) | 287 | 291 | 289
  CP: Change at Day 1, Cycle 4: Sitting SBP | 1.00 (14.60) | 0.10 (16.75) | 0.60 (15.61)
  MP/OP: Change at Day 1, Cycle 1: Sitting SBP: number analyzed (Participants) | 253 | 266 | 253
  MP/OP: Change at Day 1, Cycle 1: Sitting SBP | -1.80 (15.12) | -1.60 (16.64) | 0.00 (14.81)
  MP/OP: Change at Day 15, Cycle 1: Sitting SBP: number analyzed (Participants) | 241 | 249 | 3
  MP/OP: Change at Day 15, Cycle 1: Sitting SBP | -1.10 (14.37) | -3.20 (16.44) | -4.70 (10.21)
  MP/OP: Change at Day 29, Cycle 1: Sitting SBP: number analyzed (Participants) | 233 | 249 | 3
  MP/OP: Change at Day 29, Cycle 1: Sitting SBP | -2.20 (15.81) | -2.80 (15.93) | -9.30 (8.14)
  MP/OP: Change at Day 1, Cycle 2: Sitting SBP: number analyzed (Participants) | 229 | 247 | 226
  MP/OP: Change at Day 1, Cycle 2: Sitting SBP | -1.20 (15.16) | -0.60 (15.46) | -0.50 (14.43)
  MP/OP: Change at Day 15, Cycle 2: Sitting SBP: number analyzed (Participants) | 219 | 236 | 0
  MP/OP: Change at Day 15, Cycle 2: Sitting SBP | -2.10 (14.44) | -3.90 (16.20) |
  MP/OP: Change at Day 29, Cycle 2: Sitting SBP: number analyzed (Participants) | 215 | 225 | 0
  MP/OP: Change at Day 29, Cycle 2: Sitting SBP | -2.70 (13.79) | -2.90 (15.28) |
  Change at EOT: Sitting SBP: number analyzed (Participants) | 137 | 116 | 120
  Change at EOT: Sitting SBP | 1.70 (16.96) | -1.00 (17.56) | 2.90 (16.69)

16. Secondary Outcome: Change From Baseline in Vital Signs - Pulse Rate at Day 1 of Cycles 2, 3, 4 in Chemotherapy Phase; Days 1, 15 and 29 of Cycles 1 and 2 in Maintenance/ Observation Phase and at End of Treatment
Description: Vital signs included blood pressure and pulse rate. Changes from baseline in sitting pulse rate were summarized. MP is applicable only for two arms 'Chemotherapy followed by Avelumab' and 'Chemotherapy + Avelumab followed by Avelumab'. OP is applicable only for third arm 'Chemotherapy followed by Observation'. Category titles 'MP/OP' imply which ever phase was applicable for the respective reporting arms.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 318 | 317 | 316
beats per minute
  CP: Change at Day 1, Cycle 2: number analyzed (Participants) | 310 | 304 | 301
  CP: Change at Day 1, Cycle 2 | -0.5 (12.34) | 1.80 (12.04) | -0.70 (11.42)
  CP: Change at Day 1, Cycle 3: number analyzed (Participants) | 305 | 298 | 295
  CP: Change at Day 1, Cycle 3 | -0.20 (12.71) | 2.90 (13.64) | -0.0 (12.29)
  CP: Change at Day 1, Cycle 4: number analyzed (Participants) | 287 | 290 | 289
  CP: Change at Day 1, Cycle 4 | -0.30 (13.49) | 1.90 (13.86) | -0.30 (14.02)
  MP/OP: Change at Day 1, Cycle 1: number analyzed (Participants) | 253 | 266 | 253
  MP/OP: Change at Day 1, Cycle 1 | -1.90 (13.70) | -0.10 (13.99) | -0.70 (13.02)
  MP/OP: Change at Day 15, Cycle 1: number analyzed (Participants) | 241 | 249 | 3
  MP/OP: Change at Day 15, Cycle 1 | -2.90 (12.94) | -2.40 (13.57) | -11.70 (15.14)
  MP/OP: Change at Day 29, Cycle 1: number analyzed (Participants) | 233 | 249 | 3
  MP/OP: Change at Day 29, Cycle 1 | -3.10 (12.48) | -3.60 (13.48) | -4.00 (7.55)
  MP/OP: Change at Day 1, Cycle 2: number analyzed (Participants) | 228 | 247 | 226
  MP/OP: Change at Day 1, Cycle 2 | -3.50 (13.71) | -4.70 (13.09) | -3.40 (13.11)
  MP/OP: Change at Day 15, Cycle 2: number analyzed (Participants) | 219 | 236 | 0
  MP/OP: Change at Day 15, Cycle 2 | -5.10 (13.73) | -4.90 (13.67) |
  MP/OP: Change at Day 29, Cycle 2: number analyzed (Participants) | 215 | 225 | 0
  MP/OP: Change at Day 29, Cycle 2 | -5.60 (13.71) | -5.20 (12.79) |
  Change at EOT: number analyzed (Participants) | 136 | 116 | 119
  Change at EOT | -1.60 (14.47) | -1.50 (15.22) | -3.70 (15.03)

17. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: ECG abnormalities included: 1) QT interval, QT interval corrected using Bazett's formula (QTcB) and QT interval corrected using Fridericia's formula (QTcF): increase from baseline greater than (>) 30 millisecond (ms) or 60 ms; absolute value > 450 ms, >480 ms and > 500 ms; 2) heart rate (HR) : absolute value <=50 bpm and decrease from baseline >=20 bpm; absolute value >=120 beats per minute (bpm) and increase from baseline >=20 bpm; 3) PR interval: absolute value >=220 ms and increase from baseline >=20 ms; 4) QRS interval: absolute value >= 120 ms.
Time Frame: Baseline to discontinuation from the study or death, whichever occurred first (maximum duration of 27 months)
Population: The safety analysis set included all participants who had received at least one dose of study drug. Here "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and 'Number analyzed' = participants in the safety analysis set who had at least one baseline and post-baseline ECG assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 317 | 321 | 320
Participants
  QT increase from baseline >30 ms: number analyzed (Participants) | 314 | 314 | 314
  QT increase from baseline >30 ms | 128 | 152 | 106
  QT increase from baseline >60 ms: number analyzed (Participants) | 314 | 314 | 314
  QT increase from baseline >60 ms | 31 | 60 | 35
  QT >450 ms | 12 | 30 | 20
  QT >480 ms | 2 | 10 | 7
  QT >500 ms | 1 | 6 | 5
  QTcB increase from baseline >30 ms: number analyzed (Participants) | 300 | 303 | 306
  QTcB increase from baseline >30 ms | 107 | 137 | 116
  QTcB increase from baseline >60 ms: number analyzed (Participants) | 300 | 303 | 306
  QTcB increase from baseline >60 ms | 19 | 38 | 25
  QTcB >450 ms: number analyzed (Participants) | 303 | 312 | 313
  QTcB >450 ms | 135 | 185 | 165
  QTcB >480 ms: number analyzed (Participants) | 303 | 312 | 313
  QTcB >480 ms | 29 | 63 | 32
  QTcB >500 ms: number analyzed (Participants) | 303 | 312 | 313
  QTcB >500 ms | 16 | 29 | 17
  QTcF increase from baseline >30 ms: number analyzed (Participants) | 300 | 303 | 306
  QTcF increase from baseline >30 ms | 90 | 125 | 89
  QTcF increase from baseline >60 ms: number analyzed (Participants) | 300 | 303 | 306
  QTcF increase from baseline >60 ms | 14 | 34 | 17
  QTcF >450 ms: number analyzed (Participants) | 303 | 312 | 313
  QTcF >450 ms | 44 | 83 | 53
  QTcF >480 ms: number analyzed (Participants) | 303 | 312 | 313
  QTcF >480 ms | 10 | 25 | 15
  QTcF >500 ms: number analyzed (Participants) | 303 | 312 | 313
  QTcF >500 ms | 6 | 11 | 11
  Heart rate <=50 bpm and decrease >= 20 bpm: number analyzed (Participants) | 300 | 303 | 306
  Heart rate <=50 bpm and decrease >= 20 bpm | 1 | 1 | 3
  Heart rate >=120 bpm and increase >= 20 bpm: number analyzed (Participants) | 300 | 303 | 306
  Heart rate >=120 bpm and increase >= 20 bpm | 7 | 10 | 6
  PR >=220 ms and increase from baseline >=20 ms: number analyzed (Participants) | 312 | 311 | 313
  PR >=220 ms and increase from baseline >=20 ms | 7 | 6 | 6
  QRS >=120 ms | 7 | 9 | 16

18. Secondary Outcome: Functional Assessment of Ovarian Symptom Index- 18 (FOSI-18) Score
Description: National Comprehensive Cancer Network-Functional Assessment of Cancer Therapy (NCCN-FACT) Ovarian Symptom Index-18 (FOSI-18) is an 18-itemed participant completed questionnaire, designed to assess impact of cancer therapy on ovarian cancer-related symptoms. Based on numerical point scoring of symptoms. Includes three subscales: disease-related symptoms (10 items), treatment-related side effects (5) and general function/well-being (3). Participants rated their level of symptoms for each items using 5-point scale from 0=not at all to 4=very much. Items that were negatively framed, scores were reversed for analysis so that higher scores= good quality of life. Total symptom index: total of 18 scores, ranging from 0=severely symptomatic to 72=asymptomatic. Higher FOSI-18 scores= better functioning or lower symptom burden. MP applicable only for arms 'Chemotherapy followed by Avelumab' and 'Chemotherapy + Avelumab followed by Avelumab' and OP for 'Chemotherapy followed by Observation'.
Time Frame: CP: Pre-dose on Day 1 of Cycles 2 to 6 (1 cycle= 21 days); MP/OP: Day 1 of Cycles 1 to 12 (1 cycle= 42 days), End of treatment (any time up to Month 27)
Population: The full analysis set included all randomized participants. Here, 'Number analyzed' = participants evaluable for this outcome measure at specified rows. Category titles 'MP/OP' imply which ever phase was applicable for the respective reporting arms.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 332 | 331 | 335
units on a scale
  CP: Day 1, Cycle 2: number analyzed (Participants) | 313 | 311 | 321
  CP: Day 1, Cycle 2 | 54.33 [53.5 to 55.2] | 53.88 [53.0 to 54.7] | 54.27 [53.4 to 55.1]
  CP: Day 1, Cycle 3: number analyzed (Participants) | 312 | 311 | 317
  CP: Day 1, Cycle 3 | 54.61 [53.8 to 55.5] | 54.10 [53.2 to 54.9] | 54.51 [53.6 to 55.4]
  CP: Day 1, Cycle 4: number analyzed (Participants) | 296 | 309 | 308
  CP: Day 1, Cycle 4 | 54.88 [54.0 to 55.7] | 54.31 [53.5 to 55.1] | 54.75 [53.9 to 55.6]
  CP: Day 1, Cycle 5: number analyzed (Participants) | 292 | 300 | 303
  CP: Day 1, Cycle 5 | 55.16 [54.3 to 56.0] | 54.53 [53.7 to 55.4] | 54.99 [54.1 to 55.8]
  CP: Day 1, Cycle 6: number analyzed (Participants) | 282 | 295 | 297
  CP: Day 1, Cycle 6 | 55.43 [54.6 to 56.3] | 54.74 [53.9 to 55.6] | 55.23 [54.4 to 56.1]
  MP/OP: Day 1, Cycle 1: number analyzed (Participants) | 262 | 277 | 266
  MP/OP: Day 1, Cycle 1 | 55.70 [54.9 to 56.5] | 54.96 [54.1 to 55.8] | 55.47 [54.6 to 56.3]
  MP/OP: Day 1, Cycle 2: number analyzed (Participants) | 248 | 264 | 243
  MP/OP: Day 1, Cycle 2 | 56.25 [55.4 to 57.1] | 55.39 [54.6 to 56.2] | 55.95 [55.1 to 56.8]
  MP/OP: Day 1, Cycle 3: number analyzed (Participants) | 234 | 242 | 233
  MP/OP: Day 1, Cycle 3 | 56.80 [55.9 to 57.7] | 55.82 [55.0 to 56.7] | 56.43 [55.6 to 57.3]
  MP/OP: Day 1, Cycle 4: number analyzed (Participants) | 212 | 227 | 208
  MP/OP: Day 1, Cycle 4 | 57.35 [56.5 to 58.2] | 56.25 [55.4 to 57.1] | 56.91 [56.0 to 57.8]
  MP/OP: Day 1, Cycle 5: number analyzed (Participants) | 180 | 198 | 189
  MP/OP: Day 1, Cycle 5 | 57.90 [57.0 to 58.8] | 56.69 [55.8 to 57.6] | 57.39 [56.4 to 58.3]
  MP/OP: Day 1, Cycle 6: number analyzed (Participants) | 143 | 167 | 148
  MP/OP: Day 1, Cycle 6 | 58.45 [57.5 to 59.4] | 57.12 [56.1 to 58.1] | 57.87 [56.9 to 58.9]
  MP/OP: Day 1, Cycle 7: number analyzed (Participants) | 116 | 131 | 120
  MP/OP: Day 1, Cycle 7 | 59.00 [57.9 to 60.1] | 57.55 [56.5 to 58.6] | 58.36 [57.3 to 59.4]
  MP/OP: Day 1, Cycle 8: number analyzed (Participants) | 94 | 104 | 98
  MP/OP: Day 1, Cycle 8 | 59.55 [58.4 to 60.7] | 57.98 [56.9 to 59.1] | 58.84 [57.7 to 60.0]
  MP/OP: Day 1, Cycle 9: number analyzed (Participants) | 73 | 82 | 77
  MP/OP: Day 1, Cycle 9 | 60.09 [58.9 to 61.3] | 58.41 [57.2 to 59.6] | 59.32 [58.1 to 60.5]
  MP/OP: Day 1, Cycle 10: number analyzed (Participants) | 57 | 59 | 64
  MP/OP: Day 1, Cycle 10 | 60.64 [59.4 to 61.9] | 58.84 [57.6 to 60.1] | 59.80 [58.5 to 61.1]
  MP/OP: Day 1, Cycle 11: number analyzed (Participants) | 42 | 38 | 52
  MP/OP: Day 1, Cycle 11 | 61.19 [59.8 to 62.6] | 59.28 [57.9 to 60.6] | 60.28 [58.9 to 61.7]
  MP/OP: Day 1, Cycle 12: number analyzed (Participants) | 22 | 27 | 37
  MP/OP: Day 1, Cycle 12 | 61.74 [60.3 to 63.2] | 59.71 [58.3 to 61.1] | 60.76 [59.3 to 62.2]
  End of treatment: number analyzed (Participants) | 301 | 301 | 297
  End of treatment | 57.04 [56.2 to 57.9] | 56.01 [55.1 to 56.9] | 56.64 [55.8 to 57.5]

19. Secondary Outcome: European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Score
Description: EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). In VAS, participants rated their overall health status from 0 (worst imaginable) to 100 (best imaginable). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. Published weights are available that allow for the creation of a single summary score. 57 overall scores ranged from 0 to 1, with low scores representing a higher level of dysfunction.
Time Frame: Baseline to discontinuation from the study or death, whichever occurred first (maximum duration of 36 months)
Population: as for outcome 11
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Chemotherapy Phase: Maximum Plasma Concentration (Cmax) of Paclitaxel (Once a Week [QW] Regimen)
Description: Cmax is maximum plasma concentration of paclitaxel. The LLQ of paclitaxel was 10.0 ng/mL.
Time Frame: Pre-dose and at 1, 3, 4, 5, 6, 10, and 24 hours post paclitaxel infusion on Day 1 of Cycle 2
Population: Paclitaxel PK parameter analysis set: all participants who received at least one dose of study drug and who had at least one of the PK parameters of interest for paclitaxel. Here "Overall number of participants analyzed" signifies participants who received Paclitaxel infusion on QW regimen and had data available for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- PK: Chemotherapy Followed by Avelumab: In chemotherapy phase, participants received paclitaxel once every three weeks (Q3W) (or once weekly [QW] on Days 1, 8 and 15), followed by carboplatin Q3W on Day 1 of each 21 day cycle for 6 cycles. During the maintenance phase, participants received avelumab once every 2 weeks (Q2W) on Days 1, 15 and 29 of each 42 day cycle.
- PK: Chemotherapy + Avelumab Followed by Avelumab: In chemotherapy phase, participants received paclitaxel Q3W (or QW on Days 1, 8 and 15), followed by carboplatin Q3W along with avelumab Q3W on Day 1 of each 21 day cycle for 6 cycles. During the maintenance phase, participants received avelumab Q2W (on Days 1, 15 and 29 of each 42 day cycle).
- PK: Chemotherapy Followed by Observation: In chemotherapy phase, participants received paclitaxel Q3W (or QW on Day 1, 8 and 15), followed by carboplatin Q3W on Day 1 of each 21 day cycle for 6 cycles.
Arm/Group | PK: Chemotherapy Followed by Avelumab | PK: Chemotherapy + Avelumab Followed by Avelumab | PK: Chemotherapy Followed by Observation
Number analyzed (Participants) | 6 | 4 | 9
ng/mL | 2880 (44) | 2678 (22) | 2649 (35)

21. Secondary Outcome: Chemotherapy Phase: Maximum Plasma Concentration (Cmax) of Paclitaxel (Once Every Three Weeks [Q3W] Regimen)
Description: Cmax is maximum plasma concentration of paclitaxel. The LLQ of paclitaxel was 10.0 ng/mL.
Time Frame: Pre-dose and at 1, 3, 4, 5, 6, 10, and 24 hours post paclitaxel infusion on Day 1 of Cycle 2
Population: Paclitaxel PK parameter analysis set: all participants who had received at least one dose of study drug and who had at least one of the PK parameters of interest for paclitaxel. Here "Overall number of participants analyzed" signifies participants who received Paclitaxel infusion on Q3W regimen and had data available for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- PK: Chemotherapy Followed by Avelumab: In chemotherapy phase, participants received paclitaxel Q3W (or QW on Days 1, 8 and 15), followed by carboplatin Q3W on Day 1 of each 21 day cycle for 6 cycles. During the maintenance phase, participants received avelumab Q2W on Days 1, 15 and 29 of each 42 day cycle.
Arm/Group | PK: Chemotherapy Followed by Avelumab | PK: Chemotherapy + Avelumab Followed by Avelumab | PK: Chemotherapy Followed by Observation
Number analyzed (Participants) | 7 | 5 | 9
ng/mL | 5646 (68) | 4775 (24) | 4694 (28)

22. Secondary Outcome: Chemotherapy Phase: Maximum Plasma Concentration (Cmax) of Carboplatin (Total and Free)
Description: Cmax is maximum plasma concentration of carboplatin. The LLQ of carboplatin was 100.0 ng/mL.
Time Frame: Pre-dose and at 0.5, 1, 5, 6, 10, and 24 hours post carboplatin infusion on Day 1 of Cycle 2
Population: Carboplatin PK parameter analysis set included all participants who had received at least one dose of study drug and who had at least one of the PK parameters of interest for carboplatin. Here "Overall number of participants analyzed" signifies participants who had data available for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PK: Chemotherapy Followed by Avelumab | PK: Chemotherapy + Avelumab Followed by Avelumab | PK: Chemotherapy Followed by Observation
Number analyzed (Participants) | 11 | 7 | 13
ng/mL
  Total Carboplatin | 23580 (34) | 18350 (44) | 18990 (31)
  Free Carboplatin | 21740 (39) | 15350 (65) | 17090 (33)

23. Secondary Outcome: Chemotherapy Phase: Area Under the Plasma Concentration Time Curve From Time Zero to Infinite Time (AUCinf) of Paclitaxel (QW Regimen)
Description: AUCinf is the area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: Pre-dose and at 1, 3, 4, 5, 6, 10, and 24 hours post paclitaxel infusion on Day 1 of Cycle 2
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PK: Chemotherapy Followed by Avelumab | PK: Chemotherapy + Avelumab Followed by Avelumab | PK: Chemotherapy Followed by Observation
Number analyzed (Participants) | 5 | 4 | 7
nanogram*hour per milliliter (ng*hr/mL) | 5138 (39) | 4997 (15) | 4921 (18)

24. Secondary Outcome: Chemotherapy Phase: Area Under the Plasma Concentration Time Curve From Time Zero to Infinite Time (AUCinf) of Paclitaxel (Q3W Regimen)
Description: AUCinf is the area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: Pre-dose and at 1, 3, 4, 5, 6, 10, and 24 hours post paclitaxel infusion on Day 1 of Cycle 2
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PK: Chemotherapy Followed by Avelumab | PK: Chemotherapy + Avelumab Followed by Avelumab | PK: Chemotherapy Followed by Observation
Number analyzed (Participants) | 7 | 4 | 8
ng*hr/mL | 18070 (58) | 16190 (25) | 17470 (26)

25. Secondary Outcome: Chemotherapy Phase: Area Under the Plasma Concentration Time Curve From Time Zero to Infinite Time (AUCinf) of Carboplatin (Total and Free)
Description: AUCinf is the area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: Pre-dose and at 0.5, 1, 5, 6, 10, and 24 hours post carboplatin infusion on Day 1 of Cycle 2
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PK: Chemotherapy Followed by Avelumab | PK: Chemotherapy + Avelumab Followed by Avelumab | PK: Chemotherapy Followed by Observation
Number analyzed (Participants) | 11 | 6 | 13
ng*hr/mL
  Total Carboplatin: number analyzed (Participants) | 1 | 5 | 5
  Total Carboplatin | 87600 | 100500 (13) | 90430 (18)
  Free Carboplatin | 55840 (25) | 52000 (29) | 52300 (25)

26. Secondary Outcome: Chemotherapy Phase: Area Under the Concentration Time Curve From Time Zero to 24 Hours (AUC24) of Paclitaxel (QW Regimen)
Description: AUC24 is the area under the plasma concentration versus time curve from time zero (pre-dose) to 24 hours post-dose (0 to 24).
Time Frame: Pre-dose (0 hour), 1, 3, 4, 5, 6, 10, and 24 hours post paclitaxel infusion on Day 1 of Cycle 2
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PK: Chemotherapy Followed by Avelumab | PK: Chemotherapy + Avelumab Followed by Avelumab | PK: Chemotherapy Followed by Observation
Number analyzed (Participants) | 6 | 4 | 9
ng*hr/mL | 4960 (38) | 4572 (16) | 4304 (24)

27. Secondary Outcome: Chemotherapy Phase: Area Under the Concentration Time Curve From Time Zero to 24 Hours (AUC24) of Paclitaxel (Q3W Regimen)
Description: as for outcome 26
Time Frame: Pre-dose (0 hour), 1, 3, 4, 5, 6, 10, and 24 hours post paclitaxel infusion on Day 1 of Cycle 2
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PK: Chemotherapy Followed by Avelumab | PK: Chemotherapy + Avelumab Followed by Avelumab | PK: Chemotherapy Followed by Observation
Number analyzed (Participants) | 7 | 5 | 9
ng*hr/mL | 17540 (60) | 15870 (21) | 16390 (26)

28. Secondary Outcome: Chemotherapy Phase: Area Under the Concentration Time Curve From Time Zero to 24 Hours (AUC24) of Carboplatin (Total and Free)
Description: AUC24 is the area under the plasma concentration versus time curve from time zero (pre-dose) to 24 hours post-dose.
Time Frame: Pre-dose (0 hour), 0.5, 1, 5, 6, 10, and 24 hours post carboplatin infusion on Day 1 of Cycle 2
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PK: Chemotherapy Followed by Avelumab | PK: Chemotherapy + Avelumab Followed by Avelumab | PK: Chemotherapy Followed by Observation
Number analyzed (Participants) | 11 | 7 | 13
ng*hr/mL
  Total Carboplatin | 84380 (22) | 84100 (12) | 80960 (17)
  Free Carboplatin | 56880 (25) | 52100 (26) | 52590 (24)

29. Secondary Outcome: Maintenance Phase: Predose Plasma Concentration (Ctrough) of Avelumab
Description: Ctrough is the concentration at the end of the dosing interval when avelumab was given as a Q2W regimen in the absence of carboplatin and paclitaxel following 1 cycle of avelumab dosing, i.e. before administration of drug on Day 1 of cycle 2. Ctrough of Avelumab in the absence of chemotherapy (i.e. in the maintenance phase) has been reported. The LLQ of avelumab was 0.20 micro-gram per milliliter (mcg/mL). Data for this outcome measure was not reported for reporting arms "PK: Chemotherapy + Avelumab followed by Avelumab" (since data was not planned to be collected 1 cycle after the initiation of avelumab dosing ) and "PK: Chemotherapy followed by Observation" (since avelumab was not administered in this arm and therefore data collection was not planned).
Time Frame: Pre-dose (0 hour) on Day 1 of Cycle 2
Population: Avelumab PK concentration analysis set included all participants who had received at least one dose of study drug and who had at least one post-dose concentration measurement above the LLQ for avelumab. Here "Overall number of participants analyzed" signifies participants who had data available for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | PK: Chemotherapy Followed by Avelumab
Number analyzed (Participants) | 209
mcg/mL | 29.18 (57)

30. Secondary Outcome: Maintenance Phase: Maximum Plasma Concentration (Cmax) of Avelumab
Description: Cmax is the concentration at the end of a 1 hour infusion, corresponding to the maximum plasma concentration of avelumab. The LLQ of avelumab was 0.20 mcg/mL. Data for this outcome measure was not reported for reporting arms "PK: Chemotherapy + Avelumab followed by Avelumab"(since data was not planned to be collected 1 cycle after the initiation of avelumab dosing ) and "PK: Chemotherapy followed by Observation" (since avelumab was not administered in this arm and therefore data collection was not planned).
Time Frame: End of avelumab infusion on Day 1 of Cycle 2
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | PK: Chemotherapy Followed by Avelumab
Number analyzed (Participants) | 174
mcg/mL | 205.6 (50)

31. Secondary Outcome: Chemotherapy Phase: Maximum Plasma Concentration (Cmax) of Avelumab When Given With Paclitaxel and Carboplatin
Description: Cmax is the concentration at the end of a 1 hour infusion, corresponding to the maximum plasma concentration of avelumab. The LLQ of avelumab was 0.20 mcg/mL. Data for this outcome measure was not reported for reporting arms "PK: Chemotherapy followed by Avelumab" (data not available for this OM as avelumab was not given along with paclitaxel and carboplatin in this arm) and "PK: Chemotherapy followed by Observation" (since avelumab was not administered in this arm and therefore data collection was not planned).
Time Frame: End of infusion on Day 1 of Cycle 2
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | PK: Chemotherapy + Avelumab Followed by Avelumab
Number analyzed (Participants) | 220
mcg/mL | 162.9 (139)

32. Secondary Outcome: Chemotherapy Phase: Predose Plasma Concentration (Ctrough) of Avelumab When Given With Paclitaxel and Carboplatin
Description: Ctrough is the concentration at the end of the dosing interval when avelumab was given as a Q2W regimen in the absence of carboplatin and paclitaxel following 1 cycle of avelumab dosing, i.e. before administration of drug on Day 1 of cycle 2. The LLQ of avelumab was 0.20 mcg/mL. Data for this outcome measure was not reported for reporting arms "PK: Chemotherapy followed by Avelumab" (data not available for this OM as avelumab was not given along with paclitaxel and carboplatin in this arm) and "PK: Chemotherapy followed by Observation" (since avelumab was not administered in this arm and therefore data collection was not planned).
Time Frame: Pre-dose (0 hour) on Day 1 of Cycle 2
Population: Avelumab PK concentration analysis set included all participants who had received at least one dose of study drug and who had at least one post-dose concentration measurement above the LLQ for avelumab. Here "Overall number of participants analyzed" signifies only those participants who had data available for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | PK: Chemotherapy + Avelumab Followed by Avelumab
Number analyzed (Participants) | 251
mcg/mL | 3.607 (113)

33. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) Against Avelumab by Never and Ever Positive Status
Description: ADA against avelumab in serum samples was determined and reported separately for ADA never-positive and ADA ever-positive participants. Participants were considered ADA ever-positive if they had at least one positive (ADA titer greater than or equal to 60 with assay cut point of 1.12) ADA result at any time point during 36 months and were otherwise considered negative. Data for this outcome measure was not planned to be collected and analyzed for reporting arm "Chemotherapy followed by Observation", since, avelumab was not administered in this arm.
Time Frame: Up to 36 months
Population: The immunogenicity analysis set included all participants who had received at least one dose of study drug and who had at least one ADA sample collected for avelumab in the avelumab containing arms. Here "Overall number of participants analyzed" signifies participants who had data available for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Immunogenicity: Chemotherapy Followed by Avelumab: In chemotherapy phase, participants received paclitaxel Q3W (or QW on Days 1, 8 and 15), followed by carboplatin Q3W on Day 1 of each 21 day cycle for 6 cycles. During the maintenance phase, participants received avelumab Q2W on Days 1, 15 and 29 of each 42 day cycle.
- Immunogenicity: Chemotherapy + Avelumab Followed by Avelumab: In chemotherapy phase, participants received paclitaxel Q3W (or QW on Days 1, 8 and 15), followed by carboplatin Q3W along with avelumab Q3W on Day 1 of each 21 day cycle for 6 cycles. During the maintenance phase, participants received avelumab Q2W (on Days 1, 15 and 29 of each 42 day cycle).
Arm/Group | Immunogenicity: Chemotherapy Followed by Avelumab | Immunogenicity: Chemotherapy + Avelumab Followed by Avelumab
Number analyzed (Participants) | 272 | 328
Participants
  Never-positive | 231 | 197
  Ever-positve | 41 | 131

34. Secondary Outcome: Number of Participants With Neutralizing Antibodies (nAb) Against Avelumab by Never and Ever Positive Status
Description: nAb against avelumab in serum samples was determined and reported separately for nAb never-positive and nAb ever-positive participants. Participants were considered nAb ever-positive if they had at least one positive nAb results (less than or equal to cut point of 0.710 in qualitative competitive ligand binding assay) at any time point during 36 months. nAb never-positive participants were those who had at least one negative nAb results (greater than cut point of 0.710 in qualitative competitive ligand binding assay) at any time point. Data for this outcome measure was not planned to be collected and analyzed for reporting arm "Chemotherapy followed by Observation", since, avelumab was not administered in this arm.
Time Frame: Up to 36 months
Population: The immunogenicity analysis set included all participants who had received at least one dose of study drug and who had at least one nAb sample collected for avelumab in the avelumab containing arms. Here "Overall number of participants analyzed" signifies participants who had data available for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Immunogenicity: Chemotherapy Followed by Avelumab | Immunogenicity: Chemotherapy + Avelumab Followed by Avelumab
Number analyzed (Participants) | 272 | 328
Participants
  Never-positive | 256 | 282
  Ever-positive | 16 | 46

35. Secondary Outcome: Number of Participants With Positive Programmed Death Receptor-1 Ligand-1 (PD-L1) Biomarker Expression in Tumor Tissue as Assessed by Immunohistochemistry (IHC)
Description: PD-L1 assessment was performed using immunohistochemistry. Participants were considered positive if their pretreatment tumor tissue sample demonstrated cell surface PD-L1 expression greater than or equal to (>=) 1 percent (%) tumor cells or >= 5% immune cells and were otherwise considered negative.
Time Frame: Up to 36 months
Population: PD-L1 biomarker analysis set included all participants who had received at least one dose of study drug and who had at least one screening biomarker assessment for PD-L1.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 270 | 263 | 280
Participants | 158 | 160 | 169

36. Secondary Outcome: Number of Participants With Positive Tumor-Infiltrating Cluster of Differentiation 8 (CD8+) T Lymphocytes Expression in Tumor Tissue as Assessed by Immunohistochemistry (IHC)
Description: CD8 assessment was performed using immunohistochemistry. Participants were considered positive if their pre-treatment tumor tissue sample demonstrated >= 1% CD8 positive cells and were otherwise considered negative.
Time Frame: Up to 36 months
Population: CD8 biomarker analysis set included all participants who had received at least one dose of study drug and who had at least one screening biomarker assessment for CD8.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
Number analyzed (Participants) | 250 | 250 | 257
Participants | 107 | 107 | 118

ADVERSE EVENTS:
Time Frame: Baseline up to maximum duration of 36 months
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety set.
Arm/Group | Chemotherapy Followed by Avelumab | Chemotherapy + Avelumab Followed by Avelumab | Chemotherapy Followed by Observation
All-Cause Mortality (participants affected / at risk) | 34/328 | 31/329 | 20/334
Serious Adverse Events (participants affected / at risk) | 92/328 | 118/329 | 64/334
Other Adverse Events (participants affected / at risk) | 320/328 | 325/329 | 317/334
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy Followed by Avelumab (N=328) | Chemotherapy + Avelumab Followed by Avelumab (N=329) | Chemotherapy Followed by Observation (N=334)
Abdominal abscess (Infections and infestations) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 4
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 8 | 6
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 5 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0
Chest pain (General disorders) | 3 | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 3
Contrast media allergy (Immune system disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 1
Depression suicidal (Psychiatric disorders) | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 1
Disease progression (General disorders) | 1 | 3 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1
Embolism (Vascular disorders) | 1 | 2 | 0
Empyema (Infections and infestations) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 8 | 7
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 2 | 1 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0 | 0
Hyperpyrexia (General disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypopituitarism (Endocrine disorders) | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 3 | 4 | 9
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Incarcerated hernia (General disorders) | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infected lymphocele (Infections and infestations) | 0 | 1 | 1
Infection (Infections and infestations) | 1 | 1 | 1
Influenza (Infections and infestations) | 0 | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 4 | 0
Intestinal dilatation (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 4 | 6 | 6
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Lymph gland infection (Infections and infestations) | 1 | 0 | 0
Lymphocele (Vascular disorders) | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 5 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pelvic infection (Infections and infestations) | 0 | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 0 | 1 | 0
Perforation (General disorders) | 0 | 1 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0 | 1
Persistent depressive disorder (Psychiatric disorders) | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pneumonia (Infections and infestations) | 3 | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 3
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 2 | 0
Pyrexia (General disorders) | 6 | 10 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sarcoidosis (Immune system disorders) | 1 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 2 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 7 | 1
Subclavian vein occlusion (Vascular disorders) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 2
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 5 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 7 | 7 | 2
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Urogenital fistula (Renal and urinary disorders) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 2 | 1 | 0
Vaginal cuff dehiscence (Injury, poisoning and procedural complications) | 1 | 1 | 1
Vaginal perforation (Reproductive system and breast disorders) | 0 | 1 | 0
Viral infection (Infections and infestations) | 2 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 7 | 6
Vulval abscess (Infections and infestations) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound infection (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Essential hypertension (Vascular disorders) | 1 | 0 | 0
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy Followed by Avelumab (N=328) | Chemotherapy + Avelumab Followed by Avelumab (N=329) | Chemotherapy Followed by Observation (N=334)
Abdominal distension (Gastrointestinal disorders) | 22 | 17 | 18
Abdominal pain (Gastrointestinal disorders) | 69 | 68 | 58
Abdominal pain upper (Gastrointestinal disorders) | 32 | 39 | 24
Alanine aminotransferase increased (Investigations) | 28 | 33 | 20
Alopecia (Skin and subcutaneous tissue disorders) | 167 | 169 | 177
Anaemia (Blood and lymphatic system disorders) | 148 | 151 | 140
Anxiety (Psychiatric disorders) | 14 | 18 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 76 | 85 | 57
Aspartate aminotransferase increased (Investigations) | 18 | 28 | 21
Asthenia (General disorders) | 35 | 46 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 36 | 31
Constipation (Gastrointestinal disorders) | 113 | 100 | 95
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 55 | 22
Cystitis (Infections and infestations) | 19 | 7 | 8
Decreased appetite (Metabolism and nutrition disorders) | 64 | 55 | 37
Diarrhoea (Gastrointestinal disorders) | 84 | 101 | 63
Dizziness (Nervous system disorders) | 45 | 38 | 28
Dysgeusia (Nervous system disorders) | 22 | 20 | 18
Dyspepsia (Gastrointestinal disorders) | 31 | 24 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 38 | 47 | 29
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 12 | 12
Fatigue (General disorders) | 123 | 115 | 110
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 | 18 | 11
Headache (Nervous system disorders) | 55 | 51 | 30
Hot flush (Vascular disorders) | 23 | 18 | 16
Hypoaesthesia (Nervous system disorders) | 12 | 21 | 13
Hypokalaemia (Metabolism and nutrition disorders) | 22 | 27 | 20
Hypomagnesaemia (Metabolism and nutrition disorders) | 32 | 42 | 27
Hypothyroidism (Endocrine disorders) | 34 | 33 | 5
Infusion related reaction (Injury, poisoning and procedural complications) | 26 | 30 | 19
Insomnia (Psychiatric disorders) | 52 | 39 | 32
Leukopenia (Blood and lymphatic system disorders) | 27 | 28 | 20
Malaise (General disorders) | 22 | 17 | 14
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20 | 15 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 67 | 53 | 43
Nausea (Gastrointestinal disorders) | 153 | 149 | 152
Neuropathy peripheral (Nervous system disorders) | 63 | 77 | 65
Neutropenia (Blood and lymphatic system disorders) | 112 | 125 | 113
Neutrophil count decreased (Investigations) | 60 | 54 | 75
Oedema peripheral (General disorders) | 27 | 29 | 23
Pain (General disorders) | 21 | 23 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 30 | 32 | 37
Paraesthesia (Nervous system disorders) | 18 | 26 | 10
Peripheral sensory neuropathy (Nervous system disorders) | 91 | 76 | 82
Platelet count decreased (Investigations) | 25 | 39 | 44
Procedural pain (Injury, poisoning and procedural complications) | 27 | 22 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 38 | 37 | 19
Pyrexia (General disorders) | 33 | 42 | 23
Rash (Skin and subcutaneous tissue disorders) | 59 | 66 | 25
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 | 21 | 5
Stomatitis (Gastrointestinal disorders) | 28 | 24 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 46 | 62 | 59
Upper respiratory tract infection (Infections and infestations) | 27 | 28 | 14
Urinary tract infection (Infections and infestations) | 36 | 46 | 28
Vomiting (Gastrointestinal disorders) | 86 | 74 | 66
White blood cell count decreased (Investigations) | 32 | 31 | 34
Dry mouth (Gastrointestinal disorders) | 17 | 10 | 5
Nasopharyngitis (Infections and infestations) | 18 | 16 | 10
Weight decreased (Investigations) | 15 | 17 | 13
Hypertension (Vascular disorders) | 16 | 19 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-06-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT02718417/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT02718417/SAP_001.pdf